CLINICAL TRIAL: NCT02264080
Title: Phase I Clinical Study of WAL2014 (Talsaclidine) Capsule: A Multiple Oral Dose Study
Brief Title: Pharmacokinetics and Safety of WAL2014 (Talsaclidine) Administered Orally to Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 506.112
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — talsaclidine fumarate

ARMS (2):
- WAL2014 (Experimental)
  Interventions: Drug: WAL2014
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WAL2014
  Other Names: Talsaclidine
  Arms: WAL2014
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the pharmacokinetics and safety of WAL2014 capsules administered orally as a multiple dose to healthy adult male volunteers in double blind manner.

ELIGIBILITY:
Inclusion Criteria:

Subjects for the study are healthy male adult volunteers who meet all the inclusion criteria listed below and do not fall into the exclusion criteria.

1. Age: 20-30 years old
2. Body weight: 50-80 kg
3. Obesity index: within +/-20% of the standard body weight [standard body weight = (height - 100) x 0.9]
4. Those who have received screening examinations listed in Table 1 within one month prior to the start of the clinical study and have been judged as eligible by the investigator. Results of the simple test for gastric acidity are not used as the basis of the judgment.
5. Those who belong to volunteer members' association which has an office in Clinical Pharmacology Center, Ohsaki Clinic

Exclusion Criteria:

1. Those who have a history of allergic reaction or hypersensitivity to drugs
2. Those who have received any kind of drug(s) within one week prior to the administration of the investigational product.
3. Those who have ingested alcoholic drink within two days before the administration of the investigational product
4. Those who have been admitted to a hospital, undergone surgery or donated blood within 3 months before the administration of the investigational product
5. Those who have participated in a phase I clinical study of a drug which contains a new active ingredient or a similar study within 4 months before the administration of the investigational product
6. Those who participated in Phase I single dose study of the investigational product
7. Those who have a history of liver or renal disease
8. Those who are judged as ineligible for the clinical study by the investigator

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1999-03; Primary Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of the analyte in plasma (Cmax) | up to day 14
Time to reach maximum plasma concentration (tmax) | up to day 14
Area under the plasma concentration-time curve (AUC) | up to day 14
Urinary excretion rate | up to day 14
Minimum plasma concentration (Cmin) | up to day 14
Mean residence time (MRT) | up to day 14
Terminal half-life (t1/2) | up to day 14
Distribution volume | up to day 14
Total clearance | up to day 14
Number of subjects with adverse events | up to 22 days